CLINICAL TRIAL: NCT01495234
Title: A Pilot Investigation of Recombinant Human Bone Morphogenetic Protein- 2/Biphasic Calcium Phosphate in Patients With Spinal Degeneration With Instability Requiring Surgical Fusion
Brief Title: Pilot Study of rhBMP-2/BCP in Patients With Spinal Degeneration With Instability Requiring Surgical Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOC#1187b BCP -Mexico
Record Dates: First submitted 2011-12-12; First posted 2011-12-19 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease
Keywords: Spinal degeneration
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Each patient will receive 15mg of rhBMP-2 in rhBMP-2/BCP device and implant unilaterally during a posterolateral spinal fusion procedure. The contralateral side was fused using standard fusion techniques with autograft bone.
  Interventions: Device: rhBMP-2/BCP device
- Cohort 2 (Experimental): Each patient will receive 20mg of rhBMP-2 in rhBMP-2/BCP device and implant bilaterally.
  Interventions: Device: rhBMP-2/BCP device

INTERVENTIONS:
Device: rhBMP-2/BCP device — The rhBMP-2/BCP device consists of recombinant human Bone Morphogenetic Protein-2 (rhBMP-2) and the biphasic calcium phosphate (BCP) carrier.
  Other Names: Recombinant human bone morphogenetic protein-2
  Arms: Cohort 1
Device: rhBMP-2/BCP device — The rhBMP-2/BCP device consists of recombinant human Bone Morphogenetic Protein-2 (rhBMP-2) and the biphasic calcium phosphate (BCP) carrier.
  Other Names: recombinant human Bone Morphogenetic Protein-2
  Arms: Cohort 2

SUMMARY:
This study is designed to generate data relating to patient safety, bone generating activity associated with the use of the rhBMP-2/BCP device as compared to autograft and to evaluate the feasibility of conducting a larger clinical trial in a patient population requiring spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Subject has radiographically documented spinal degeneration with instability as documented by the presence of translation >= 4mm or angulation >= 5°.
* Subject has intractable back pain which does not respond to conservative treatment and in the investigator's opinion, requires surgical spinal fusion.
* Subject's pain is predominantly associated with the back.
* Subject has only one level involvement at L3-L4, L4-L5, or L5-S1.
* Subject is 18 years of age or greater at the time consent is given to participate in the study.
* Subject is willing to comply with the study plan and sign the informed consent.
* Subject is male or a non-pregnant, non-nursing female. All females of child-bearing age must agree to use adequate contraception for a period of no less than 16 weeks following surgery.

Exclusion Criteria:

* Subject has primary spinal diagnosis of a disorder other than spinal degeneration with instability at the involved surgical level.
* Subject has spinal stenosis or condition which requires a full laminectomy procedure.
* Subject has had a previous fusion, discectomy or laminectomy procedure at L3-L4, L4-L5 or L5-S1.
* Subject has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids, methotrexate) or has a condition which requires postoperative medications that interfere with fusion (e.g., steroids, nonsteroidal antiinflammatory drugs, or methotrexate).
* Subject has overt or active infection near the operative spinal region.
* Subject has active systemic infection.
* Subject has history of autoimmune disease (Systemic Lupus Erythematosus or Dermatomyositis).
* Subject's history includes hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins).
* Subject has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/BCP implantation.
* The subject requires electrical bone growth stimulation, allograft, or bone substitute as part of treatment.
* Subject has history of endocrine or metabolic disorder known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, Ehlers Danlos syndrome, or osteogenesis imperfecta).
* Subject has a known diagnosis of diabetes which requires treatment with medication.
* Subject has received previous radiation therapy at the site to be fused.
* Subject is unwilling to return for required follow-up visits.
* Subject is a prisoner.
* Subject has insufficient bone mass which precludes surgery (e.g., severe osteopenia or osteoporosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1996-10; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Fusion Status | 12 month
  Fusion will be met all of the following criteria:
  1. Evidence of bridging trabecular bone;
  2. Angular motion < 5°;
  3. Translational motion <= 3mm;
  4. No radiolucent lines spanning the entire fusion mass.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Disability Questionnaire Status | 12 month
Neuro/Functional Status | 12 month
  A neurological functional questionnaire will be completed by patients prior to surgery and postoperative, including three questions pertaining to pain (severity of pain, location of pain, and leg pain side), and four questions associated with functional activities (recreational activity level, putting on shoes and socks, squatting, occupation activity level). Success will be based on a maintenance or improvement from the preoperative condition for the functional components, except that severity of pain success will be based on an improvement of at least one point on the five point scale.
Neurological Status | 12 month
  A scale will be used to measure neurological status. This scale focuses on reflexes, sensory, motor function, and the degree of straight leg raise reproducing pain. All of these elements are combined to give an overall score. Success will be based on a maintenance or improvement in all categories from the preoperative condition.
General Health Status (SF-36) | 12 month